CLINICAL TRIAL: NCT04849026
Title: A Randomized, Open Label, Multiple-dose, 2-way Crossover, Phase I Study to Compare the Safety and Pharmacokinetics Profile of WID-CLZ18 and Clozaril 100 mg Tablet (Clozapine) After Oral Administration in Schizophrenia Patients
Brief Title: Bioequivalence Study in Patients With Schizophrenia by Using Clozaril 100 mg Tablet (Clozapine) and WID-CLZ18
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Whanin Pharmaceutical Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: WID-CLZ18-BE
Record Dates: First submitted 2021-04-14; First posted 2021-04-19 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Clozapine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Experimental): 1. Period 1: WID-CLZ18
  2. Period 2: Clozaril 100 mg (Clozapine)
  Interventions: Drug: Clozaril 100 mg (Clozapine); Drug: WID-CLZ18
- Group B (Experimental): 1. Period 1: Clozaril 100 mg (Clozapine)
  2. Period 2: WID-CLZ18
  Interventions: Drug: Clozaril 100 mg (Clozapine); Drug: WID-CLZ18

INTERVENTIONS:
Drug: Clozaril 100 mg (Clozapine) — 2 Doses/Day for 10 days
Drug: WID-CLZ18 — 2 Doses/Day for 10 days

SUMMARY:
This clinical study is a randomized, open label, multiple-dose, 2-way crossover, phase I (Bioequivalence) study to compare the safety and pharmacokinetics profile of WID-CLZ18 and Clozaril 100 mg tablet (Clozapine) after oral administration in schizophrenia patients.

ELIGIBILITY:
Main Inclusion Criteria:

1. Males and females adults aged 20 to 65 years
2. Diagnosed as schizophrenia prior to the screening visit
3. On treatment with a stable dose of clozapine 200 mg/day for at least 12 weeks before the screening visit and taken at 100 mg twice daily during the study period

Main Exclusion Criteria:

1. Subjects who have a medical history specified in protocol
2. Subjects with confirmed abnormal laboratory values specified in protocol
3. Subjects who have a medication history or safety risks specified in protocol
4. Subjects who can not comply with requirements of pharmacokinetic sampling as per protocol
5. Subjects who are expected to have the prohibited concomitant medication therapy during the study period
6. Pregnant women or breast-feeding women or men and women who has possibility of pregnancy
7. Subjects who are not suitable for the clinical trial

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-08-14 (Actual)

PRIMARY OUTCOMES:
Cmax | Up to 12 hours
  Maximum blood concentration in steady state
AUC0-12 | Up to 12 hours
  Area under the concentration-time curve from zero to 12 hours at steady state

SECONDARY OUTCOMES:
Tmax | Up to 12 hours
  Time to maximum blood concentration
T1/2 | Up to 12 hours
  Terminal elimination half life
R | Up to 12 hours
  Accumulation rate
Cmin | Up to 12 hours
  Steady-state peak plasma concentration
Fluctuation | Up to 12 hours
  (Cmax-Cmin)/Cav

CONTACTS AND LOCATIONS:
Overall Officials: Bo-Hyun Yoon, Principal Investigator — Department of Psychiatry, Naju National Hospital
Locations (1):
- Whan In Pharm., Seoul, South Korea